CLINICAL TRIAL: NCT05695937
Title: Effect of the Adapted Brazilian Cardioprotective Diet Supplemented With Phytosterols and/or Krill Oil in Patients With Familial Hypercholesterolemia: DICA-HF Pilot Study
Brief Title: Brazilian Cardioprotective Diet, Phytosterols and Krill Oil in Patients With Familial Hypercholesterolemia
Acronym: DICA-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: University of Sao Paulo (Other); National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DICA-HF_PILOT
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Phytosterols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DICA-HF + placebo (Placebo Comparator): Participants allocated into this arm (n= 24) will receive the DICA Br adapted to FH (DICA-HF) plus placebo of both phytosterol and krill oil during 120 days.
  Interventions: Other: Placebo phytosterol; Other: Placebo krill oil
- DICA-HF + phytosterol (Experimental): Participants allocated into this arm (n= 24) will receive the DICA Br adapted to FH (DICA-HF) plus 2g/day of phytosterol and placebo of the krill oil during 120 days.
  Interventions: Dietary Supplement: phytosterol; Other: Placebo krill oil
- DICA-HF + krill oil (Experimental): Participants allocated into this arm (n= 24) will receive the DICA Br adapted to FH (DICA-HF) plus 2g/day of krill oil and placebo of phytosterol during 120 days.
  Interventions: Dietary Supplement: krill oil; Other: Placebo phytosterol
- DICA-HF + phytosterol + krill oil (Experimental): Participants allocated into this arm (n= 24) will receive the DICA Br adapted to FH (DICA-HF) plus 2g/day of phytosterol and 2g/day of krill oil during 120 days.
  Interventions: Dietary Supplement: phytosterol; Dietary Supplement: krill oil

INTERVENTIONS:
Dietary Supplement: phytosterol — 2g/day will be provided to the participants, aiming to guarantee a minimum of 800mg/day of free phytosterols.
  Arms: DICA-HF + phytosterol; DICA-HF + phytosterol + krill oil
Dietary Supplement: krill oil — 2g/day will be provided to the participants, aiming to guarantee a minimum of 400mg/day of eicosapentaenoic (EPA) and docosahexaenoic (DHA) fatty acids.
  Arms: DICA-HF + krill oil; DICA-HF + phytosterol + krill oil
Other: Placebo phytosterol — Placebo of phytosterol, in the same quantity of the active phytosterol
  Arms: DICA-HF + krill oil; DICA-HF + placebo
Other: Placebo krill oil — Placebo of krill oil, in the same quantity of the active krill oil
  Arms: DICA-HF + phytosterol; DICA-HF + placebo

SUMMARY:
The main objective of this pilot study is to evaluate the effects of the Brazilian Cardioprotective Diet (DICA Br) supplemented or not with phytosterols and/or krill oil in patients with a probable or definitive diagnosis of familial hypercholesterolemia (FH) identified by the Dutch Lipid Clinic Network (Dutch MEDPED) criteria. In addition, the following will be considered secondary objectives: to perform participants´ complete sequencing of the exome; to evaluate the effects of the interventions on lipid profile; to identify subclasses of low-density lipoprotein (LDL) and high-density lipoprotein (HDL) cholesterol; to perform untargeted lipidomic analyses; to evaluate the frequency of mild, moderate and severe adverse events according to study groups; and to evaluate both implementation components and adherence rates to the protocol, aiming to design a larger randomized trial. In this pilot study, between 48 and 76 individuals will be randomly enrolled into four groups: 1) DICA Br adapted to FH (DICA-HF) + phytosterol placebo + krill oil placebo (control group); 2) DICA-HF + 2g/day of phytosterol + krill oil placebo; 3) DICA-HF + phytosterol placebo + 2g/day of krill oil; and 4) DICA-HF + 2g/day of phytosterol + 2g/day of krill oil. Primary outcomes will be LDL-cholesterol for groups phytosterol vs. placebo and lipoprotein(a) for groups krill oil vs. placebo after 120 days of follow up.

World Health Organization Universal Trial Number (WHO-UTN): U1111-1296-7102

DETAILED DESCRIPTION:
DICA-HF pilot study is a superiority, factorial, and in parallel randomized placebo-controlled (double-dummy) clinical trial. The randomization will be in blocks of varying sizes stratified by research center, and the allocation ratio will be 1:1:1:1. Participants will come from at least 9 center sites in different Brazilian geographic regions.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (age ≥20 years);
* Definitive (certainty) or probable diagnosis of FH by the Dutch MEDPED criteria;
* Using one of the following treatment regimens for ≥ 6 weeks: simvastatin 40 mg; lovastatin 40 mg; pravastatin 80 mg; atorvastatin 20 mg; rosuvastatin 10 mg; pitavastatin 4 mg; fluvastatin 80 mg; atorvastatin 40 - 80 mg; rosuvastatin 20 - 40 mg; atorvastatin 40 - 80 mg + ezetimibe 10mg; rosuvastatin 20 - 40 mg + ezetimibe 10mg; or simvastatin 40mg + ezetimibe 10mg.

Exclusion Criteria:

* "Possible" diagnosis of FH according to the Dutch MEDPED criteria;
* Fasting triglycerides ≥ 500mg/dL;
* Diagnosis of hypercholesterolemia due to a secondary cause (hypothyroidism, nephrotic syndrome, etc.);
* Food allergies (food, dyes, preservatives);
* Contraindication to the use of phytosterols (for example: diagnosis of sitosterolemia);
* HIV positive in treatment/AIDS;
* Chronic inflammatory diseases;
* Liver disease or chronic kidney disease on dialysis;
* Cancer under treatment or life expectancy < 6 months;
* Episode of acute coronary syndrome in the last 60 days;
* Chemical dependency/alcoholism;
* Chronic use of anti-inflammatory, anticonvulsant and immunosuppressive drugs;
* Use of PCSK9 inhibitors (alirocumab and evolocumab);
* Pregnancy or lactation;
* Wheelchair users unable to undergo anthropometric assessment;
* Body mass index ≥40kg/m²;
* Use of dietary supplements that may interfere with the outcomes of interest;
* Participation in other randomized clinical trials;
* Refusal to participate in the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
LDL-c | 120 days
  Low-density lipoprotein cholesterol, in mg/dL
Lp(a) | 120 days
  Lipoprotein(a), in mg/dL
Adherence | 120 days
  Adherence to treatment, evaluated by: attendance at consultations (at least 3 of the 4 planned study visits); plasma concentrations of phytosterols and erythrocyte levels of EPA/DHA fatty acids (identified by the difference between the last and the first study visits); and counting the consumed products under investigation (consumption of at least 80% of the capsules provided to the participants, regardless of the allocation group).

SECONDARY OUTCOMES:
TC | 120 days
  Total cholesterol, in mg/dL
HDL-c | 120 days
  High density lipoprotein cholesterol, in mg/dL
TG | 120 days
  Fasting triglycerides, in mg/dL
VLDL | 120 days
  Very low-density lipoprotein cholesterol, in mg/dL
NHDL | 120 days
  Non-HDL cholesterol, in mg/dL, calculated according to the mathematical formula: CT - HDL-c
CI I | 120 days
  Castelli Index I, in mg/dL, calculated according to the mathematical formula: CT/HDL-c
CI II | 120 days
  Castelli Index II, in mg/dL, calculated according to the mathematical formula: LDL-c/HDL-c
TG/HDL-c | 120 days
  TG/HDL-c ratio, in mg/dL, calculated according to the mathematical formula: TG/HDL-c
AI | 120 days
  Atherogenic index, in mg/dL, calculated according to the mathematical formula: NHDL/HDL-c
ox-LDL | 120 days
  Oxidized LDL, in µg/mL
AE | 120 days
  Adverse events (mild, moderate and severe), registered as percentage per study group
Implementation | 120 days
  Implementation components, measured by: on-time recruitment rates; choice and adjustments of remote platform/media for center sites training; measures of participants´ engagement to interventions; and rates of loss to follow-up.

OTHER OUTCOMES:
Subfractions | 120 days
  Subclasses of LDL-c and HDL-c, in mg/dL
Lipidomics | 120 days
  Analyses of untargeted lipidomic (all lipid species will be expressed in mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Aline Marcadenti, PhD, Principal Investigator — Hospital do Coracao; Adriana B Carvalho, PhD, Study Chair — Instituto Nacional de Cardiologia; Alexandre B Cavalcanti, PhD, Study Chair — Hospital do Coracao; Angela C Bersch-Ferreira, PhD, Study Chair — Real e Benemérita Associação Portuguesa de Beneficência; Elizabeth S Torres, PhD, Study Chair — University of Sao Paulo; Erlon O Abreu-Silva, MSc, Study Chair — Hospital do Coracao; Geni R Sampaio, PhD, Study Chair — University of Sao Paulo; Julia P Krey, RDN, Study Chair — Hospital do Coracao; Karina L Negrelli, DVM, Study Chair — Hospital do Coracao; Luis Gustavo S Mota, RDN, Study Chair — Hospital do Coracao; Marcelo M Rogero, PhD, Study Chair — University of Sao Paulo; Maria Cristina Izar, PhD, Study Chair — Universidade Federal de São Paulo; Nagila T Damasceno, PhD, Study Chair — University of Sao Paulo; Patrícia V de Luca, MSc, Study Chair — Associação Brasileira de Hipercolesterolemia Familiar; Pedro M Barros, PhD, Study Chair — Hospital do Coracao; Renato N Santos, Stat, Study Chair — Hospital do Coracao; Rosana Perim, MSc, Study Chair — Hospital do Coracao; Thaís Martins, MD, Study Chair — Hospital de Clínicas de Porto Alegre
Locations (9):
- Brazil (9):
  - Hospital São José, Criciúma
  - Hospital das Clínicas da Universidade Federal de Goiás, Goiânia
  - Universidade Regional do Noroeste do Estado do Rio Grande do Sul, Ijuí
  - Instituto Nacional de Cardiologia, Rio de Janeiro
  - Hospital Ana Nery, Salvador
  - Universidade Feevale, São Leopoldo
  - Hcor, São Paulo
  - InCor, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided